CLINICAL TRIAL: NCT03686813
Title: Sildenafil for Prevention of Swimming-Induced Pulmonary Edema (SIPE)
Brief Title: Sildenafil for Swimming-Induced Pulmonary Edema (SIPE) Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00100971
Record Dates: First submitted 2018-09-24; First posted 2018-09-27 (Actual); Results first posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-10

CONDITIONS: Edema, Pulmonary; Immersion; Diving
MeSH Terms: conditions — Pulmonary Edema | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Double blind, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Each participant will be studied with active drug and placebo.
  Interventions: Drug: Placebo Oral Tablet
- Sildenafil (Active Comparator): Sildenafil 50 mg orally one hour (once) before immersed exercise
  Interventions: Drug: Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil Citrate — Oral sildenafil, 50 mg
  Other Names: Viagra; Revatio
  Arms: Sildenafil
Drug: Placebo Oral Tablet — Placebo
  Arms: Placebo

SUMMARY:
This trial is testing the effectiveness of a single oral dose of sildenafil (50 mg) taken 1 hour before a provocative event on the subsequent development of swimming-induced pulmonary edema.

DETAILED DESCRIPTION:
Immersion pulmonary edema (also known as swimming-induced pulmonary edema, SIPE) is a condition in which the lungs fill with fluid (pulmonary edema) during a dive or vigorous swim, causing cough with bloody sputum, shortness of breath and reduced blood oxygen levels. In the Navy this usually occurs in young, healthy individuals such as SEAL and Special Warfare Combatant-Craft trainees. SIPE generally resolves spontaneously within 24 hours but it can be fatal. It is believed that SIPE is responsible for some deaths in civilians during triathlons. This proposal aims to test a drug to prevent SIPE.

Depending upon severity, the prevalence of SIPE is reported in up to 60% during 2.4-3.6 km open sea swimming trials in the Israel Defense Force. In SEAL training in the US approximately 40 cases per year (around 3%) have been reported, more commonly during winter, when it is observed in up to 5% of trainees. Return to duty time can be up to 7 days. SIPE also affects other groups of highly fit individuals such as triathletes. In susceptible individuals it tends to recur, thus a preventive medicine would be useful for both Navy SEALs and civilians.

The aim of this study will be to provide the Navy an FDA-approved drug that can be used to prevent SIPE. The investigators hypothesize that sildenafil administration to SIPE-susceptible individuals one hour before a swim in cold water will reduce or eliminate the risk of SIPE. The method to be used to test this hypothesis will be a 40-minute period of exercise immersed to the neck in 20°C water, a test that results in SIPE symptoms in the majority of susceptible individuals. The investigators plan to study 20 individuals who have previously experienced SIPE. Each volunteer will be tested twice. Either sildenafil or an inactive drug (placebo) administered in random order will be given prior to each exercise. For each participant exercise periods will be performed at least 7 days apart. The identity of the drug and placebo will be concealed from the investigators and the volunteers until the end of the study. The number of instances in which SIPE manifestations after sildenafil and placebo will then be compared.

Availability of a drug that can prevent SIPE would provide the Navy with a useful tool that could be administered to SEALs who have experienced SIPE prior to critical missions. It would also be useful for civilians who have experienced SIPE but wish to continue with the precipitating exercise such as swimming or competing in triathlons, and also for patients with heart failure for whom swimming induces shortness of breath or pulmonary edema.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 18 and 45 years
* History of swimming-induced pulmonary edema

Exclusion Criteria:

* Pregnant women
* Significant heart valve disease
* Cardiomyopathy
* Uncontrolled hypertension
* Coronary artery disease
* Obstructive lung disease
* VO2max <25 mL/kg as estimated by the University of Houston Non-Exercise Test
* Previous adverse reaction to sildenafil
* Use of antihypertensives or other drugs that are known to interact adversely with sildenafil (e.g. nitrates, alpha adrenergic blockers)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be published in the open literature

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Oral Tablet, Then Sildenafil Citrate: Each participant first received placebo oral tablet one hour (once) before immersed exercise. After a washout period of at least 7 days, they then received Sildenafil citrate 50 mg orally one hour (once) before immersed exercise.
- Sildenafil Citrate, Then Placebo Oral Tablet: Each participant first received Sildenafil citrate 50 mg orally one hour (once) before immersed exercise. After a washout period of at least 7 days, they then received placebo oral tablet one hour (once) before immersed exercise.
Period: Overall Study
Arm/Group | Placebo Oral Tablet, Then Sildenafil Citrate | Sildenafil Citrate, Then Placebo Oral Tablet
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Oral Tablet, Then Sildenafil Citrate | Sildenafil Citrate, Then Placebo Oral Tablet | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (6.0) | 37.5 (6.0) | 38.1 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 8 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pulmonary Edema
Description: One or more of: hypoxemia, productive cough, pulmonary edema on chest radiograph, wheezing on chest auscultation.
Time Frame: During or immediately after exercise in cold water, approximately one hour and 40 minutes
Population: Each participant was studied with active drug and placebo.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Oral Tablet: Each participant will be studied with active drug and placebo.
  Placebo Oral Tablet: Placebo
- Sildenafil Citrate: Sildenafil 50 mg orally one hour (once) before immersed exercise
  Sildenafil Citrate: Oral sildenafil, 50 mg
Arm/Group | Placebo Oral Tablet | Sildenafil Citrate
Number analyzed (Participants) | 18 | 18
Participants | 7 | 9
Statistical Analysis 1: Comparison: Placebo Oral Tablet vs Sildenafil Citrate; Test type: Other; p = 0.317, McNemar

2. Secondary Outcome: Number of Participants With Dyspnea Leading to Voluntary Premature Cessation of Exercise
Description: Voluntary premature cessation of exercise due to shortness of breath.
Time Frame: During or immediately after exercise in cold water, approximately one hour and 40 minutes
Population: Each participant was studied with active drug and placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Oral Tablet | Sildenafil Citrate
Number analyzed (Participants) | 18 | 18
Participants | 10 | 8
Statistical Analysis 1: Comparison: Placebo Oral Tablet vs Sildenafil Citrate; Test type: Other; p = 0.317, McNemar

3. Secondary Outcome: Number of Participants With Post-exercise 10% Decrease in Forced Vital Capacity (FVC) or Forced Expiratory Volume in One Second (FEV1) as Measured by Spirometry
Description: Post-exercise 10% decrease in forced vital capacity (FVC) or forced expiratory volume in one second (FEV1).
Time Frame: Immediately after exercise in cold water, approximately one hour and 40 minutes
Population: Each participant was studied with active drug and placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Oral Tablet | Sildenafil Citrate
Number analyzed (Participants) | 18 | 18
Participants | 3 | 3
Statistical Analysis 1: Comparison: Placebo Oral Tablet vs Sildenafil Citrate; Test type: Other; p > 0.999, McNemar

4. Secondary Outcome: Number of Participants With "Comet Tails" Seen on Ultrasound of the Lungs
Description: A "comet tail" artefact is a short path reverberation artefact that weakens with each reverberation, resulting in a vertical echogenic artefact that rapidly fades as it continues in to the ultrasound image.
Time Frame: Immediately after exercise in cold water, approximately one hour and 40 minutes
Population: Each participant was studied with active drug and placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Oral Tablet | Sildenafil Citrate
Number analyzed (Participants) | 18 | 18
Participants | 17 | 14
Statistical Analysis 1: Comparison: Placebo Oral Tablet vs Sildenafil Citrate; Test type: Other; p = 0.18, McNemar

5. Secondary Outcome: Number of Participants Who Found the Exercise Easiest When Given Sildenafil Citrate Versus When Given Placebo
Time Frame: Immediately after exercise in cold water, approximately one hour and 40 minutes
Population: Each participant was studied with active drug and placebo.
Measure: Count of Participants; unit: Participants
Groups:
- Sildenafil Citrate and Placebo Oral Tablet: Each participant will be studied with active drug and placebo. Each participant first received either active drug or placebo one hour (once) before immersed exercise. After a washout period of at least 7 days, they then received the remaining option one hour (once) before immersed exercise.
Arm/Group | Sildenafil Citrate and Placebo Oral Tablet
Number analyzed (Participants) | 18
Participants
  Placebo Oral Tablet | 5
  Sildenafil Citrate | 9
  No Difference | 4
Statistical Analysis 1: Comparison: Sildenafil Citrate and Placebo Oral Tablet; Test type: Other; p = 0.29, McNemar

ADVERSE EVENTS:
Time Frame: During and immediately after exercise in cold water
Arm/Group | Placebo Oral Tablet, Then Sildenafil Citrate | Sildenafil Citrate, Then Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT03686813/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT03686813/ICF_000.pdf